CLINICAL TRIAL: NCT07388966
Title: Prospective Longitudinal Monocentric Study to Measure Limb Movement in Patients With FGFR3-related Skeletal Dysplasia Using Syde®
Brief Title: Prospective Longitudinal Monocentric Study to Measure Limb Movement in Patients With FGFR3-related Skeletal Dysplasia
Acronym: SKY-MOT3
Status: Not yet recruiting | Type: Observational
Sponsor: SYSNAV (Industry)
Responsible Party: Sponsor
Other Study IDs: PR5030-108; 2025-A01608-41 (Other: ANSM)
Record Dates: First submitted 2026-01-28; First posted 2026-02-05 (Actual); Last update posted 2026-02-05 (Actual); Status verified 2026-01

CONDITIONS: Achondroplasia; Hypochondroplasia
MeSH Terms: conditions — Achondroplasia; Hypochondroplasia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The study aims to identify which Syde®-derived digital outcomes are reliable in FGFR3-related Skeletal Dysplasia. This requires to set-up a natural history study to measure limb movements in patients with ACH or HCH.

ELIGIBILITY:
Inclusion Criteria:

1. Aged 3 years old or older at the time of consent.
2. Written informed consent obtained:

   1. From the parent(s) or legal guardian(s) for participants under 18 years old.
   2. From participants 18 years old and older.
3. Affiliated to, or beneficiary of a social security category
4. Able to walk unassisted for at least 10 meters.
5. Genetically confirmed diagnosis with one pathogenic variant (ACMG class IV & V) of achondroplasia or hypochondroplasia.
6. Participant (and caregivers for participants under 18 years old) willing and able to comply with all study procedures including: questionnaires, Syde® related procedures

Exclusion Criteria:

1. Subjects who have short stature condition other than ACH/HCH.
2. Presence of cognitive disorders that limit their understanding of the data collection process (training of device use and 4-week recording periods every 6 months, device return at the end of the study), the implication of the study and consent.
3. Presence or history of any concurrent disease or condition that could interfere with study participation, impact pediatric growth, affect motor or balance or gait function (such as neurological, endocrine, infectious, allergic, osteoarthritis, or inflammatory), assessed by the investigator.
4. Females who are pregnant, or planning to become pregnant during the study duration.
5. Body Mass Index = 35 kg/m2.
6. Recent upper and/or lower limbs injury (trauma/fracture or surgery) in the 6 months preceding inclusion.
7. Prior limb lengthening surgery or planned or expected to have limb lengthening surgery while enrolled in the study.
8. Presence of guided growth hardware (such as 8-plates) or planned orthopedic surgeries during the study.
9. Vulnerable patient (guardianship, curatorship or safeguarding of justice), unable to provide informed consent or who is unable to express their consent.

Ages: 3 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Participants will be recruited from the patient registry of the Centre de Référence des Maladies Osseuses Constitutionnelles located at NeckerHospital / IMAGINE Institute. The APPT association (Association des Personnes de Petite Taille) will also help with the recruitment through flyers distribution. All visits will take place at Necker Hospital.
Sampling Method: Non-Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2026-02 (Estimated); Primary Completion 2028-02 (Estimated); Study Completion 2028-02 (Estimated)

PRIMARY OUTCOMES:
Reliability of digital endpoint derived from Syde® assessed by the Intra-Class Correlation (ICC) for each recording period timepoint. | 12 months
  reliability assessed by the ICC (Intra-Class Correlation)for each recording period timepoint (baseline, 6 months, 12 months)

SECONDARY OUTCOMES:
number of participants reaching 180 hours of recording during the recording periods defined in the protocol | 12 months
  Number of patients reaching 180 hours of recordings during the recording periods defined in the protocol (supposed optimal threshold for Syde®-derived digital endpoint computation) at baseline, 6 months, 12 months
F-SUS (French System Usability Score) score at 6 months of Syde® use | 6 months
  F-SUS score at 6 months
Correlation between digital endpoints derived from Syde® and 6-minutes walk test (6MWT) | 12 months
  Correlation at baseline and at different timepoints between Syde® derived digital endpoint and 6MWT
Correlation between digital endpoints derived from Syde® and growth parameters | 12 months
  Correlation at baseline and at different timepoints between Syde® derived digital endpoints and annualized growth velocity, height Z-score, body proportion ratios
Correlation between digital endpoints derived from Syde® and Patient-reported Outcomes (PROs) | 12 months
  Correlation at baseline and at different timepoints between Syde® derived digital endpoints and PROs
Longitudinal Change in digital endpoints derived from Syde® | 12 months
  Change from baseline in digital endpoints derived from Syde® at 6 and 12 months
Accuracy of Syde® movement detection | Baseline
  Accuracy of Syde® movement detection compared to Optical Motion Capture measures
Qualitative interview exploring limitations on mobility and impact on daily life | baseline
  caregiver and/or participant qualitative interview exploring limitations on mobility daily life

CONTACTS AND LOCATIONS:
Overall Officials: Genevieve Baujat, Principal Investigator — Hopital Necker
Locations (1):
- Hopital Necker, Paris, France